CLINICAL TRIAL: NCT05224050
Title: Open Trial of Heart Rate Variability Biofeedback for Smoking Cessation Treatment
Brief Title: Heart Rate Variability Biofeedback for Smoking Cessation Treatment
Acronym: HRVB-SCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Teresa M. Leyro, Ph.D., Principal Investigator, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2019001539; 5R34DA043751-03 (NIH)
Record Dates: First submitted 2021-12-13; First posted 2022-02-04 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Tobacco Smoking
Keywords: Smoking Cessation; Heart Rate Variability Biofeedback
MeSH Terms: conditions — Tobacco Smoking; Smoking Cessation | interventions — Cognitive Behavioral Therapy; Biofeedback, Psychology; Tobacco Use Cessation Devices; Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: All participants will receive individualized smoking cessation therapy (SCT), nicotine replacement therapy patch (NRT) and heart rate variability biofeedback (HRVB)
Masking Description: This is an open trial with all participants receiving the experimental intervention (HRVB) in addition to smoking cessation therapy and nicotine replacement therapy patch.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Heart Rate Variability Biofeedback-Smoking Cessation Therapy (HRVB-SCT) (Experimental): All participants in this open trial will receive individualized training in resonance breathing using biofeedback to help improve self-regulation (HRVB), cognitive-behavioral smoking cessation treatment (SCT), and up to 8-weeks of the transdermal nicotine patch (NRT).
  Interventions: Behavioral: Cognitive-Behavioral Smoking Cessation; Biological: Heart Rate Variability Biofeedback; Drug: Nicotine patch

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Smoking Cessation — Participants will be provided with six individualized smoking cessation counseling sessions designed to help them prepare to quit, set a quit date, behaviorally manage early abstinence, and to resume cessation upon lapse.
  Other Names: Cognitive-behavioral therapy; Smoking cessation counseling
Biological: Heart Rate Variability Biofeedback — Participants will be provided with seven individualized trainings in resonance breathing using biofeedback to help improve self-regulation.
  Other Names: Biofeedback; Respiratory biofeedback
Drug: Nicotine patch — All participants will be offered up to eight weeks of transdermal nicotine patch, beginning on their quit date.
  Other Names: Transdermal nicotine patch; Nicotine replacement therapy

SUMMARY:
The purpose of the study is to conduct an open trial examining the feasibility and acceptability of an adapted heart rate variability biofeedback and smoking cessation treatment that was using a primarily virtual remote intervention.

DETAILED DESCRIPTION:
The present investigation is an open trial investigating the feasibility and acceptability of heart rate variability biofeedback smoking cessation treatment (HRVB-SCT) for individuals who smoke cigarettes. Significant findings will also support the expansion of HRVB as a transdiagnostic treatment adjunct that alters cardiac vagal functioning to promote emotional and behavioral regulation, changing the status quo of cognitive-behavioral intervention approaches and decreasing the health and economic burden of smokers who suffer from emotional distress.

The goals are to: (a) assess the feasibility and acceptability of the HRVB-SCT intervention (b) assess the efficacy of the intervention in modifying smoking behavior and emotional distress; and (c) collect additional information to inform a subsequent randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-50
* Smoking ≥ 5 cigarettes, daily, for at least two years
* Expired carbon monoxide analysis of breath sample ≥8 ppm
* A score of > 5 on the Readiness to Quit Ladder (i.e., desire to quit smoking within the next 6 months)
* Ability to read and speak English fluently
* Computer and Smartphone proficient

Exclusion Criteria:

* Use of other tobacco or nicotine products for recreation or to aid in cessation or use of medication to aid in smoking cessation or currently receiving counseling for smoking cessation
* Endorsement of current or past psychotic or manic symptoms indicative of bipolar spectrum or schizophrenia spectrum disorders and/or current suicidal or homicidal ideation
* Self-reported pending legal issue with potential to result in incarceration
* Plan to move from the New Brunswick, New Jersey area within the next 6 months
* Inability to provide written informed consent
* Current evidence of another substance use disorder
* Severe visual or hearing impairments
* Self-reported medical condition or medication use that may be contraindicated for participation in heart rate variability biofeedback training or confound autonomic parameters: Being overweight or obese (i.e., body mass index > 35); Severe asthma or breathing problems (e.g., chronic obstructive pulmonary disease, emphysema, bronchitis); currently pregnant or lactating or plans to become pregnant in the next 4 months; Autoimmune disorder (e.g., multiple sclerosis; under or overactive thyroid); Neurodegenerative disorder (e.g., Alzheimer's disease, Parkinson's disease); Current use of a psychotropic medication or use of other medication that may affect the cardiovascular system (e.g., mood stabilizers, anti-psychotics, monoamine oxidase inhibitors, tricyclics, beta blockers, benzodiazepines; patients taking selective serotonin reuptake inhibitors or selective norepinephrine reuptake inhibitors will be enrolled if on a stable regimen for at least 6 weeks); History of heart murmur or arrhythmia; Pacemaker or other implanted cardiac devices; Heart disease; or Abnormal heart or respiratory parameters including respiration rate > 20 breaths per minute, extra systoles, or hypertension (e.g., blood pressure reading ≥ 140/90; this may be determined following baseline assessment. Importantly, the presence of any of these exclusion factors, if unknown to the participant would not put them at any risk if they participated in the study, it would simply make the cardiovascular data more difficult (if not impossible) to process and interpret, and
* Self-reported medical issues of potential concern to nicotine patch users (i.e., unstable angina pectoris, myocardial infarction, or significant cardiac arrhythmia (including atrial fibrillation) in the past 90 days

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa M, Leyro, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers, School of Arts and Sciences, One Spring Street, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leyro TM, Buckman JF, Bates ME. Theoretical implications and clinical support for heart rate variability biofeedback for substance use disorders. Curr Opin Psychol. 2019 Dec;30:92-97. doi: 10.1016/j.copsyc.2019.03.008. Epub 2019 Apr 2. PMID 31055246

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the greater Rutgers, New Brunswick community via posters, leaflets, mailings, online advertisements, community outreach (i.e., meetings with local organizations and treatment providers), and listservs. The first participant was enrolled 11/29/2021 and the last participant was enrolled 03/15/2023.
Pre-assignment Details: The intervention involved 7 sessions (2 in-person and 5 virtual remote) scheduled over a 6-week period. All participants received individualized heart rate variability biofeedback at each session, smoking cessation therapy during 6 of the sessions, and 8 weeks of transdermal nicotine patches.
Groups:
- Heart Rate Variability Biofeedback-Smoking Cessation Therapy (HRVB-SCT): All participants in this open trial received individualized heart rate variability biofeedback training (HRVB), cognitive-behavioral smoking cessation treatment (SCT), and up to 8-weeks of the transdermal nicotine patch (NRT).
  Heart Rate Variability Biofeedback: Participants were provided with seven individualized trainings in resonance breathing using biofeedback to help improve self-regulation.
  Cognitive-Behavioral Smoking Cessation: Participants were provided with six individualized smoking cessation counseling sessions designed to help them prepare to quit, set a quit date, behaviorally manage early abstinence, and to resume cessation upon lapse.
  Nicotine patch: Participants were offered up to eight weeks of transdermal nicotine patch, beginning on their quit date.
Period: Overall Study
Arm/Group | Heart Rate Variability Biofeedback-Smoking Cessation Therapy (HRVB-SCT)
Started | 28
Treatment Completed | 19
Follow-up Completed | 16
Completed | 16
Not Completed | 12
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Groups:
- Enrolled: Participants who were eligible and completed the Baseline session
Arm/Group | Enrolled
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 18
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility: Participant Attendance
Description: Number of intervention sessions attended out of 7 possible sessions.
Time Frame: 6 weeks
Population: Data on the Intent-to-treat N=28 participants who completed the baseline session and were enrolled in the study.
Measure: Mean (Standard Deviation); unit: Sessions
Groups:
- Intent-to-treat Sample: Participants who completed their baseline session, enrolled, and completed at least one session of the intervention.
Arm/Group | Intent-to-treat Sample
Number analyzed (Participants) | 28
Sessions | 5.32 (2.28)

2. Primary Outcome: Intervention Feasibility: Participant Practice Adherence
Description: Time (in minutes) spent practicing the breathing intervention
Time Frame: 6 weeks
Population: Data on the Intent-to-treat N=28 participants who completed the baseline session and were enrolled in the study.
Measure: Mean (Standard Deviation); unit: Minutes per day
Arm/Group | Intent-to-treat Sample
Number analyzed (Participants) | 28
Minutes per day | 8.01 (6.03)

3. Primary Outcome: Intervention Feasibility: Participant Ratings of Effectiveness
Description: Effectiveness was assessed via self-report ratings on four items assessing the intervention in terms of helping them quit and manage emotional distress, rated on a 0=completely disagree to 4=completely agree Likert-type scale. Mean total scores were computed by averaging the items for each respective timepoint. Mean total scores range from 0-4. For this scale, higher scores are indicative of greater perceived intervention efficacy.
Time Frame: Week 1 (i.e., treatment initiation), Week 6 (i.e., end of treatment/1-month post-quit), and Week 16 (i.e., 3-MFU)
Population: Of the N=28 participants who enrolled in the study, n=27 had available data at Week 1 for this measure; Of the n=19 who completed treatment, n=18 had data available at Week 6; n=16 completed this measure at their 3-month follow up.
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Week 1 (Treatment Initiation): Participants who enrolled and attended their first intervention session.
- Week 6 (End of Treatment): Participants who attended their 1-Month Post-Quit session.
- Week 16 (3-MFU): Participants who attended their 3-month follow up session.
Arm/Group | Week 1 (Treatment Initiation) | Week 6 (End of Treatment) | Week 16 (3-MFU)
Number analyzed (Participants) | 27 | 18 | 16
score on scale | 3.02 (0.59) | 3.29 (0.59) | 2.80 (0.90)

4. Primary Outcome: Intervention Feasibility: Participant Ratings of Appropriateness
Description: Appropriateness was assessed via self-report ratings on two items assessing the intervention in terms of comprehension and fit, rated on a 0=completely disagree to 4=completely agree Likert-type scale. Mean total scores were computed by averaging the items for each respective timepoint. Mean total scores range from 0-4. For this scale, higher scores are indicative of greater perceived intervention appropriateness.
Time Frame: Week 1 (i.e., treatment initiation), Week 6 (i.e., end of treatment/1-month post-quit), and Week 16 (i.e., 3-MFU)
Population: Of the N=28 participants who enrolled in the study, n=26 had available data at Week 1 for this measure; Of the n=19 who completed treatment, n=17 had available data at Week 6; n=16 completed this measure at their 3-month follow up.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Week 1 (Treatment Initiation) | Week 6 (End of Treatment) | Week 16 (3-MFU)
Number analyzed (Participants) | 26 | 17 | 16
score on scale | 3.46 (0.51) | 3.68 (0.47) | 3.28 (0.73)

5. Primary Outcome: Intervention Feasibility: Participant Ratings of Ease of the Intervention
Description: Ease of the Intervention was assessed via self-report ratings on three items assessing ease of use and fit into daily lifestyle, rated on a 0=completely disagree to 4=completely agree Likert-type scale. Mean total scores were computed by averaging the items for each respective timepoint. Mean total scores range from 0-4. For this scale, higher scores are indicative of greater perceived ease of the intervention and fit into daily lifestyle.
Time Frame: Week 1 (i.e., treatment initiation), Week 6 (i.e., end of treatment/1-month post-quit) and Week 16 (i.e., 3-MFU)
Population: Of the N=28 participants who enrolled in the study, n=27 had available data at Week 1 for this measure; Of the n=19 who completed treatment, n=18 had available data at Week 6; n=16 completed this measure at their 3-month follow up.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Week 1 (Treatment Initiation) | Week 6 (End of Treatment) | Week 16 (3-MFU)
Number analyzed (Participants) | 27 | 18 | 16
score on scale | 2.70 (0.58) | 2.58 (0.51) | 2.73 (0.65)

6. Primary Outcome: Intervention Feasibility: Interventionist Ratings of Technical Issues
Description: The intervention used several pieces of technology, including remote session delivery via Zoom, smartphone assisted carbon monoxide (CO) monitor and HRVB devices, remote survey administration, as well as in-person use of biofeedback and physiological monitoring equipment. Technological limitations were assessed via self-report items documenting incidences of technical issues during intervention sessions and their related effects on intervention delivery. Items include Yes/No and open-text responses.
Time Frame: 6 weeks
Population: There was a total of 291 intervention sessions where instances of technical issues could have occurred and been reported.
Measure: Number; unit: sessions with 1 or more technical issues
Units Other Than Participants: Sessions
Groups:
- Interventionist Reports of Technical Issues: Total number of intervention sessions where Interventionists could have experienced and reported technical issues
Arm/Group | Interventionist Reports of Technical Issues
Number analyzed (Participants) | NA
Number analyzed (Sessions) | 291
sessions with 1 or more technical issues | 117

7. Primary Outcome: Intervention Acceptability: Participant Rating of Satisfaction and Liking
Description: Satisfaction and liking will be assessed via self-report items regarding satisfaction with learning the intervention, liking the intervention, breathing techniques, nicotine replacement, and recommending the intervention to others. Items are rated on a 0=completely disagree to 4=completely agree Likert-type scale. Mean total scores were computed by averaging the items for each respective timepoint. Mean total scores range from 0-4. For this scale, higher scores are indicative of greater satisfaction and liking of the intervention and greater perceived intervention acceptability.
Time Frame: Week 1 (i.e., treatment initiation), Week 6 (i.e., end of treatment/1-month post-quit) and Week 16 (i.e., 3-MFU)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Week 1 (Treatment Initiation) | Week 6 (End of Treatment) | Week 16 (3-MFU)
Number analyzed (Participants) | 27 | 18 | 16
score on scale | 3.24 (0.56) | 3.68 (0.33) | 3.45 (0.62)

8. Secondary Outcome: Changes in Total Emotional Distress
Description: Self-reported change in emotional distress was evaluated via the 21-item, Depression, Anxiety and Stress Scale (DASS-21). The DASS-21 is composed of three self-report scales that measure the emotional states of depression, anxiety and stress. Items are rated on a Likert-type scale (0=Did not apply to me at all, to 3=Applied to me very much, or most of the time). Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items. The severity ratings are as follows Depression: Normal 0-4, Mild: 5-6, Moderate: 7-10, Severe: 11-13, Extremely Severe: 14-21. Anxiety: Normal: 0-3, Mild: 4-5, Moderate: 6-7, Severe: 8-9, Extremely Severe: 10-21. Stress: Normal: 0-7, Mild: 8-9, Moderate: 10-12, Severe: 13-16, Extremely Severe: 17-21. Total scores are computed by summing the subscales. Total scores for the DASS-21 range from 0-63. For all scales, higher scores are indicative of greater emotional distress and less change in total distress symptoms over time.
Time Frame: Week 0, Week 5, Week 6, and Week 16 (i.e., Baseline, 2-weeks Post-Quit, 1-Month Post-Quit, 3-MFU)
Population: Of the N=28 participants who were eligible and attended their baseline session, n=20, n=19, and n=16 attended and completed this measure at their 2-weeks post-quit, 1-month post-quit, and 3-month follow up sessions.
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Baseline: Participants who attended their baseline visit
- 2-Weeks Post-Quit: Participants who attended their 2-weeks Post-Quit session.
- 1-Month Post-Quit: Participants who attended their 1-month Post-Quit session.
- 3-MFU: Participants who attended their 3-month follow up session.
Arm/Group | Baseline | 2-Weeks Post-Quit | 1-Month Post-Quit | 3-MFU
Number analyzed (Participants) | 28 | 20 | 19 | 16
score on scale
  DASS-21 Total score | 12.50 (9.76) | 15.44 (7.38) | 18.16 (10.68) | 21.50 (11.70)
  DASS-21 Depression score | 3.39 (3.28) | 3.15 (2.82) | 4.89 (4.18) | 7.06 (4.36)
  DASS-21 Anxiety score | 3.57 (3.67) | 4.80 (2.63) | 5.11 (3.26) | 5.69 (4.09)
  DASS-21 Stress score | 5.54 (4.48) | 7.49 (3.42) | 8.16 (4.66) | 8.75 (4.85)
Statistical Analysis 1: Comparison: Baseline vs 2-Weeks Post-Quit; Test type: Other — A paired-samples t-test was conducted to examine differences in the DASS-21 total score from baseline to 2-weeks post-quit; p = 0.40, t-test, 2 sided — The threshold for statistical significance was p<0.05; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-6.98 to 2.89], Standard Deviation 10.54 — Mean difference represents the difference of the mean for the DASS-21 total scores at Baseline and at 2-weeks post-quit. The reported estimated value is based on data from the n=20 who attended their 2-weeks post-quit session
Statistical Analysis 2: Comparison: 2-Weeks Post-Quit vs 1-Month Post-Quit; Test type: Other — A paired-samples t-test was conducted to examine the difference in the DASS-21 total scores from 2-weeks post-quit to 1-month post-quit; p = 0.26, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = -2.43, 95% CI 2-sided [-6.84 to 1.98], Standard Deviation 9.15 — Mean difference represents the difference of mean DASS-21 total scores at 2-weeks post-quit and 1-month post-quit. The reported estimated value is based on data from the n=19 participants who attended their 1-month post-quit session
Statistical Analysis 3: Comparison: 1-Month Post-Quit vs 3-MFU; Test type: Other — A paired-samples t-test was conducted to examine the difference in the DASS-21 total scores from 1-month post-quit to 3-month follow up; p = 0.11, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = -2.75, 95% CI 2-sided [-6.21 to 0.71], Standard Deviation 6.49 — Mean difference represents the difference of mean DASS-21 total scores at 1-month post-quit and 3-month follow up. The reported estimated value is based on data from the n=16 participants who attended their 3-month follow up session

9. Secondary Outcome: Changes in Smoking Behavior: Quit Day Abstinence
Description: Quit day abstinence was assessed via self-reported smoking abstinence on Quit Day and verified via carbon monoxide (CO) analysis of breath sample (CO < 8ppm).
Time Frame: Week 3 (i.e., Quit Date)
Population: Of the N=28 who were eligible and initiated treatment, n=22 attended their quit date.
Measure: Count of Participants; unit: Participants
Groups:
- Quit Date: Participants who attended their Quit day session
Arm/Group | Quit Date
Number analyzed (Participants) | 22
Participants | 8

10. Secondary Outcome: Changes in Smoking Behavior: Sustained Smoking Cessation
Description: Sustained smoking cessation was assessed via self-reported abstinence at 3-months post-quit) and verified via carbon monoxide (CO) analysis (CO < 8ppm) and salivary cotinine levels (<10 ng/mL).
Time Frame: Week 16 (i.e., 3-MFU)
Population: Of the N=28 who were eligible and initiated treatment, n=16 attended their 3-month follow-up session.
Measure: Count of Participants; unit: Participants
Groups:
- 3-Month Follow Up: Participants who attended their 3-month follow-up session.
Arm/Group | 3-Month Follow Up
Number analyzed (Participants) | 16
Participants | 3

11. Secondary Outcome: Changes in Smoking Behavior: Reduced Smoking Rate
Description: Cigarettes smoked per day (CPD) assessed via self-report responses on the Timeline Followback interview were used to measure changes in smoking behavior from Baseline through Quit Date, 2-weeks post-quit, 1-month post-quit, and 3-months follow up.
Time Frame: Week 0, Week 3, Week 5, Week 6, and Week 16 (i.e., Baseline, Quit Date, 2-Weeks Post-Quit, 1-Month Post-Quit, 3-Month follow up)
Population: Of the N=28 participants who were eligible and attended their baseline session, n=22 attended their quit date, n=20 attended their 2-weeks post-quit session, n=19 attended their 1-month post-quit session, and n=16 attended their 3-month follow up.
Measure: Mean (Standard Deviation); unit: Cigarettes smoked per day (CPD)
Groups:
- Baseline: Mean CPD at baseline was determined by averaging the total number of cigarettes smoked per day for the 28 days prior to the participant's baseline session. Data reflect participants who attended their baseline session and enrolled in the study.
- Quit Date: Mean CPD at Quit date was determined by averaging the total number of cigarettes smoked on their Quit-day session. Data reflect participants who attended their Quit-day session.
- 2-Weeks Post-Quit: Mean CPD at 2-Weeks Post-Quit was determined by averaging the total number of cigarettes smoked per day for the 7 days prior to the participant's 2-weeks post-quit session. Data reflect participants who attended their 2-weeks post-quit session.
- 1-Month Post-Quit: Mean CPD at 1-Month Post-Quit was determined by averaging the total number of cigarettes smoked per day for the 7 days prior to the participant's 1-month post-quit session. Data reflect participants who attended their 1-month post-quit session.
- 3-Month Follow Up: Mean CPD at 3-Month Follow-Up was determined by averaging the total number of cigarettes smoked per day for the 7 days prior to the participant's 3MFU session. Data reflect participants who attended their 3MFU session.
Arm/Group | Baseline | Quit Date | 2-Weeks Post-Quit | 1-Month Post-Quit | 3-Month Follow Up
Number analyzed (Participants) | 28 | 22 | 20 | 19 | 16
Cigarettes smoked per day (CPD) | 14.73 (7.09) | 1.14 (2.77) | 1.09 (2.00) | 1.12 (2.80) | 3.30 (3.67)
Statistical Analysis 1: Comparison: Baseline vs Quit Date; Test type: Other — A paired-samples t-test was conducted to compare changes in cigarettes smoked per day from Baseline to Quit Day; p < 0.001, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 13.70, 95% CI 2-sided [9.88 to 17.53], Standard Deviation 8.63 — Mean difference represents the average difference in cigarettes smoked per day from Baseline to Quit Date. The reported estimated value is based on data from the n=22 participants who attended their Quit Date session
Statistical Analysis 2: Comparison: Quit Date vs 2-Weeks Post-Quit; Test type: Other — A paired-samples t-test was used to evaluate smoking reduction in participants from Quit Date to 2-weeks Post-Quit; p = 0.80, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.83 to 1.06], Standard Deviation 2.02 — Mean difference represents the average difference in cigarettes smoked per day from Quit Date to 2-weeks Post-Quit. The reported estimated value is based on data from the n=20 participants who attended their 2-weeks post-quit session
Statistical Analysis 3: Comparison: 2-Weeks Post-Quit vs 1-Month Post-Quit; Test type: Other — A paired-samples t-test was used to evaluate smoking reduction in participants from 2-weeks post-quit to 1=month post-quit; p = 0.97, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-1.41 to 1.45], Standard Deviation 2.97 — Mean difference represents the average difference in cigarettes smoked per day from 2-weeks post-quit to 1-month post-quit. The reported estimated value is based on data from the n=19 participants who attended their 1-month post-quit session
Statistical Analysis 4: Comparison: 1-Month Post-Quit vs 3-Month Follow Up; Test type: Other — A paired-samples t-test was used to evaluate smoking reduction in participants from 1-month post-quit to 3-month follow-up; p = 0.04, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = -2.17, 95% CI 2-sided [-4.17 to -0.17], Standard Deviation 3.75 — Mean difference represents the average difference in cigarettes smoked per day from 1-month post-quit to 3-month follow-up. The reported estimated value is based on data from the n=16 participants who attended their 3-month follow-up session

ADVERSE EVENTS:
Time Frame: Baseline (i.e., Week 0), End-of-Treatment (i.e., Week 6, 1-month post-quit), 2-Month Follow Up (i.e., Week 16, 3-months post-quit).
Groups:
- Heart Rate Variability Biofeedback-Smoking Cessation Therapy (HRVB-SCT): All participants in this open trial received individualized training in resonance breathing using biofeedback to help improve self-regulation (HRVB), cognitive-behavioral smoking cessation treatment (SCT), and up to 8-weeks of the transdermal nicotine patch (NRT).
  Cognitive-Behavioral Smoking Cessation: Participants was provided with six individualized smoking cessation counseling sessions designed to help them prepare to quit, set a quit date, behaviorally manage early abstinence, and to resume cessation upon lapse.
  Heart Rate Variability Biofeedback: Participants was provided with seven individualized trainings in resonance breathing using biofeedback to help improve self-regulation.
  Nicotine patch: All participants were offered up to eight weeks of transdermal nicotine patch, beginning on their quit date.
Arm/Group | Heart Rate Variability Biofeedback-Smoking Cessation Therapy (HRVB-SCT)
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT05224050/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT05224050/ICF_001.pdf